CLINICAL TRIAL: NCT04024085
Title: Time to be Ready to Void: a New Tool to Assess the Time Needed to Perform Micturition for Patients With Multiple Sclerosis
Brief Title: Time to be Ready to Void: a New Tool to Assess the Time Needed to Perform Micturition in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GRC-001 GREEN
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Gait Disorders, Neurologic; Urinary Incontinence, Urge; Multiple Sclerosis
MeSH Terms: conditions — Gait Disorders, Neurologic; Urinary Incontinence, Urge; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: adult with a multiple sclerosis diagnosis, able to walk 50 meters without human help, Expanded Disability Status Scale (EDSS) < 7, consulting in a neuro-urology department
  Interventions: Other: completion of the test created Time to be Ready to Void

INTERVENTIONS:
Other: completion of the test created Time to be Ready to Void — completion of the test created (Time to be Ready to Void) The participants have to stand up from a chair with armrests, walk 6 meters to the toilet, open the door and turn on the light, close the door, undress and position themselves to urinate

SUMMARY:
The aim of the study is to create a specific test to assess the global time required to go to the toilet and to perform micturition, at the moment the patient decides to urinate in multiple sclerosis population, and to assess its reliability.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) are frequent in central nervous system disorders especially in patients with multiple sclerosis (PwMS). Prevalence of LUTS is important (32 to 96.8%) and increases with the multiple sclerosis (MS) duration and the severity of the neurological deficiencies and disabilities. Overactive bladder with urgency, frequency, urge incontinence, is the most common symptom, reported by 37-99% of the PwMS. OAB not only impacts quality of life but overactive detrusor associated with detrusor sphincter dyssynergia can lead to upper urinary tract alteration (reflux, dilatation, urinary tract infection). In the absence of risk factor, the treatment aims to improve comfort and quality of life. Anticholinergic drugs are usually the first-line treatment, but their frequent adverse effects (constipation, xerostomia, cognitive impairment) may impact compliance and adherence. The warning time (defined as the time between the first desire to void and the micturition impossible to defer) only partially reflects the possibilities of continence. Indeed, other numerous and various factors such as patient mobility, autonomy for transfers, speed of undressing, etc., can influence the global time between the first alert (first desire to void) and the imperious micturition and thus on the risk of incontinence.

The global time required to go to the toilet and undress is difficult to quantify and no specific and validated test is available for this.

The aim of the study is to create a specific test to assess the global time required to go to the toilet and to perform micturition, at the moment the patient decides to urinate in multiple sclerosis population, and to assess its reliability.

In this study, the investigators develop a new tool to assess the global time required to go to the toilet until patients are ready to void: Time to be Ready to Void (TRV). The different stages to go to the toilet are individualized, and two prior steps are defined: a mobility stage starting when the examiner gives the starting signal, includes the stand up, the walk to the toilets, and stops when the patient puts his hand on the door handle; and a settled stage starting as soon as the subject has his hand on the door handle, until he is undressed and in his usual and secure position to void. The "interval" or "lap" function of the chronometer is used to facilitate the recording. Difficulty of each stage is assessed by a 4-point Likert type scale with 3 indicating ''no difficulty'' and 0 indicating ''impossible or necessitate human help".

This study was approved by the local ethics review board RCB: 2018-A01644-51. Participants will be recruited in a Neuro-urology department during a medical appointment, an urodynamic assessment, or a day hospital related to urinary disorders.

Data collected are:

* Medical history
* Age
* Sex
* EDSS score
* Urinary Symptom Profile score
* Data of the last urodynamic
* need to void with numerical scale between 0 and 10 before the test

To assess inter-rater reliability, two examiners record the first TRV try with both a digital chronometer. To assess reliability of the TRV, a second try is done after at least 10 minutes of rest, with one of the two examiners, checking that the need to void has not changed significantly.

To assess the internal consistency of the TRV, further tests are carried out:

* a 10-meter walk test (10MWT) at maximum speed
* a Timed Up and Go (TUG)
* a Tinetti Mobility Test
* the self-questionnaire Fall Efficacy Scale International for balance evaluation
* a bilateral Nine Hold Peg (NHP) Test for dexterity
* the Functional Independence Measure (FIM) score
* the Katz - activities of daily living index (Katz ADL)

Statistical analyses will be performed with the R software for Windows (Rx64 3.2.3, R Foundation for Statistical Computing, Vienna, Austria). Descriptive data will be presented as means with SD for continuous data and as medians with range for ordinal data and data not normally distributed.

Inter-rater reliability and test-re test reliability will be assessed using intra-class correlation coefficient (ICC, absolute agreement). Internal consistency with the complementary tests will be assessed using Spearman correlation.

ELIGIBILITY:
Inclusion Criteria:

* adult with a multiple sclerosis diagnosis,
* able to walk 50 meters without human help,
* Expanded Disability Status Scale (EDSS) < 7

Exclusion Criteria:

* relapse of multiple sclerosis in the last 7-days,
* acute urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with multiple sclerosis who were consulting in neuro-urology department
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Total time for TRV | 1 day
  The participants have to stand up from a chair with armrests, walk 6 meters to the toilet, open the door and turn on the light, close the door, undress and position themselves to urinate. All the test is timed

SECONDARY OUTCOMES:
Time for the first stage: "mobility" stage | 1 day
  , the "mobility" stage, starting when the examiner gives the starting signal, includes the stand up, the walk to the toilets, and stops when the patient puts his hand on the door handle
Time for the second stage: "settled" stage | 1 day
  the "settled" stage starts as soon as the subject has his hand on the door handle, until he is undressed and in his usual and secure position to void

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided